CLINICAL TRIAL: NCT07031102
Title: RISKA: Respiratory Irritability With School Kids With/Without Asthma - Assessment of Methacholine Responsiveness in Pediatric Asthma: A Comparative Study With Healthy Controls
Brief Title: Methacholine Challenge Test in School Children With/Without Asthma RISKA
Acronym: RISKA
Status: Recruiting | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Janne Burman, PhD, MD, Pediatric Allergist, Helsinki University Central Hospital
Other Study IDs: HUS/5351/2024
Record Dates: First submitted 2025-05-30; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Asthma Bronchiale; Lung Function Tests; Bronchial Hyperresponsiveness
Keywords: Asthma; Lung function test; children; Methacholine challange test; Bronchial provocation test
MeSH Terms: conditions — Bronchial Hyperreactivity; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controlled Asthma: Children with asthma without need to intensify asthma treatment
- Unocontrolled Asthma: Children with asthma and need to intensify their asthma treatment
- Controlls: Children without asthmatic symptoms and medication

SUMMARY:
The study includes a pre-study telephone interview with healthy controls to assess their eligibility for participation. During the study visit, a background information form and an asthma questionnaire are completed. At the study visit, a methacholine challenge test measuring airway hyperresponsiveness and an exhaled nitric oxide measurement are performed. The effect of medication intensification in asthma patients is further assessed through a telephone interview 1-2 months after the medication adjustment.

DETAILED DESCRIPTION:
Study type: Observational study Study sites: Skin and Allergy Hospital, Helsinki, Finland Inclusion criteria: Age 7-15 years, diagnosed with asthma and on regular asthma medication with physician-assessed good asthma control (55 participants), suboptimal asthma control (55 participants), or healthy controls with no inhaled asthma medication or asthma-related symptoms in the preceding two years (150 participants).

Exclusion criteria: Other respiratory, cardiovascular, or neurological diseases; acute respiratory infection within 2 weeks; respiratory disorders related to prematurity; implanted or external active medical devices.

Sample size: 110 asthma patients and 150 healthy controls. Study duration: Until the end of 2027 Study visits: One study visit; in addition, consent will be sought to contact participants during the 15-year storage period of the study data, for example, regarding questionnaire follow-ups.

Objectives:

Primary:

To determine whether airway hyperresponsiveness differs clinically significantly (PD20FEV1 at least twofold difference) between children with well-controlled asthma, those requiring intensified asthma medication, and healthy controls.

To determine whether a corresponding difference exists in exhaled nitric oxide levels between the groups.

Secondary:

To assess how age correlates with airway hyperresponsiveness (PD20FEV1 value) in the methacholine challenge among healthy controls.

To assess how sensitization to airborne allergens correlates with PD20FEV1 values in healthy controls and asthma patients.

To assess how blood eosinophil levels correlate with PD20FEV1 values in the methacholine challenge in both healthy controls and asthma patients.

Implementation:

Healthy controls will undergo a pre-study telephone interview to assess eligibility. At the study visit, background information and asthma questionnaires will be completed. The study visit will include a methacholine challenge test measuring airway hyperresponsiveness and an exhaled nitric oxide measurement. The effect of medication intensification in asthma patients will be evaluated via a telephone interview 1-2 months after the medication adjustment.

ELIGIBILITY:
Inclusion Criteria: Healthy Controls

* • Aged 7-15 years, both sexes

  * No diagnosis of asthma in childhood
  * No inhaled asthma medication during the previous 2 years
  * No wheezing or shortness of breath during the previous 2 years
  * Written informed consent from the participant and guardian

Inclusion Criteria: Children with Asthma

* Aged 7-15 years, both sexes
* Physician-diagnosed asthma (ICD-10 codes J45.0/J45.1/J45.9)
* Inhaled corticosteroid treatment for at least 6 months
* Either:

  * Well-controlled asthma (c-ACT/ACT score ≥20) and no clinical need to intensify medication, or
  * Poorly controlled asthma with physician-confirmed need for intensified asthma medication

Exclusion Criteria:

* • Premature birth before 32 gestational weeks

  * Other chronic cardiopulmonary or neurological conditions affecting airways (excluding asthma)
  * Severe underlying illness such as malignancy
  * Beta-blocker medication
  * Active immunological disease

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants:
  * 55 children with well-controlled asthma
  * 55 children with asthma symptoms despite regular asthma medication
  * 150 healthy controls without asthma symptoms in the past two years
  Recruitment:
  * Symptomatic asthma patients will be recruited from the Pediatric Allergy Unit at the Skin and Allergy Hospital, Helsinki, Finland.
  * Healthy controls will be recruited through sports clubs and schools in the Uusimaa Region, Finland
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
BHR and asthma balance | Baseline
  To determine whether airway hyperresponsiveness (defined as cumulative dose of methacholine causing 20% fall of FEV1 (PD20FEV1)) differs clinically significantly (PD20FEV1 at least twofold difference) between children with well-controlled asthma, those requiring intensified asthma medication, and healthy controls
FeNO in study groups | Baseline
  To determine whether a corresponding difference exists in exhaled nitric oxide levels between the groups

SECONDARY OUTCOMES:
Age and BHR | Baseline
  assess how age correlates with airway hyperresponsiveness (PD20FEV1 value) in the methacholine challenge among healthy controls
Allergic sensitization and BHR | Baseline
  assess how sensitization to airborne allergens correlates with PD20FEV1 values in healthy controls and asthma patients
Eosinophils and BHR | Baseline
  assess how blood eosinophil levels (absolute count) correlate with PD20FEV1 values in the methacholine challenge in both healthy controls and asthma patients

CONTACTS AND LOCATIONS:
Overall Officials: Mika Mäkelä, Professor, PhD, MD, Study Chair — HUS
Locations (1):
- HUS Skin and Allergy Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided